CLINICAL TRIAL: NCT04718766
Title: The Reliability and Validity of the Turkish Version of the Occupational Sitting and Physical Activity Questionnaire in Office Workers
Brief Title: The Reliability and Validity of the Turkish Version of the Occupational Sitting and Physical Activity Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Saime Nilay Arman, Saime Nilay ARMAN, Istanbul University - Cerrahpasa
Other Study IDs: 11971
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Physical Activity; Office Worker; Sedentary Behavior
Keywords: Physical Activity; Office Worker; Sedentary Behavior
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is to investigate the validity and reliability of the Occupational Sitting And Physical Activity Questionnaire (OSPAQ) scale in Turkish by making a cultural adaptation in office workers, which was developed to evaluate work-related sitting, standing, walking and doing heavy work. 100 office workers will be included in the study. Physical activity level of office workers will be evaluated with Turkish OSPAQ and International Physical Activity Questionnaire.

DETAILED DESCRIPTION:
It is reported that those who do desk work in working life act less as a result of their professional requirements. Considering the benefits of physical activity, it is recommended that the risks of desk workers, especially those in the risk group who produce work by consuming less energy, should be reduced and encouraged to participate in physical activity at a level and manner suitable for a healthier life. For this reason, it is important to determine the level of physical activity according to different variables in individuals working at desk jobs.The aim of our study is to evaluate the validity and reliability of the "Occupational Sitting And Physical Activity Questionnaire (OSPAQ)" scale in Turkish, which was developed to evaluate the situation of sitting, standing, walking and doing heavy work. All forms will be sent through the media. 100 office workers will be included in the study. Physical activity level of office workers will be evaluated by Turkish OSPAQ and International Physical Activity Questionnaire. For the reliability study, after 7 days, the physical activity of office workers will be re-evaluated with Turkish OSPAQ. Factor analysis methods will be used to examine the factor structure of the scale, correlation analysis (Pearson and Spearman coefficients) in validity analysis and test-retest reliability. Cronbach alpha analysis will be used in the reliability analysis.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 20-45 Being resident in Turkey Working at a desk job for at least one year Using a computer for at least 4-5 hours a day at work Volunteering to participate in the study

Exclusion Criteria:

* Exercising regularly for the last 2 months Having a cardiac, neurological or rheumatic chronic disease Being pregnant

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1000 office workers residing in Turkey will be contacted via e-mail and social media. Participants who agree to participate in the study via Google forms will be able to answer the questions. The individuals who volunteers and meets the inclusion criteria will be included in the study. at least 100 office workers will be included in the present study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-30 (Estimated); Primary Completion 2021-02-25 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
"Occupational Sitting And Physical Activity Questionnaire (OSPAQ)'' | Change from baseline to 7 day
  The OSPAQ is a brief instrument to record the proportion of work time spent sitting, standing, walking, and doing heavy labour, as well as the total length of time worked in the past five working days. Participants will be asked to indicate the percentage of time spent on those activities during working hours on a typical working day. The participants will be received a slightly adjusted instruction to fill in the OSPAQ compared to other studies, namely to keep in mind a typical working day instead of the last seven working days (i.e. "How would you describe a typical working day in your current job? This only includes your working day. Commuting and everything outside the work setting is not included."). So when accumulating all percentages a total percentage of 100 was obtained: for example, 55% occupational sitting, 25% walking, 15% standing, and 5% performing heavy labour.
International physical activity questionnaire short form | Change from baseline to 7 day
  The IPAQ has since become the most widely used physical activity questionnaire, with two versions available: the 31 item long form (IPAQ-LF) and the 9 item short form (IPAQ-SF). The short form records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting. The original authors recommended the "last 7 day recall" version of the IPAQ-SF for physical activity surveillance studies, in part because the burden on participants to report their activity is small.